CLINICAL TRIAL: NCT02363543
Title: Comparison of Hyalomatrix and Integra Wound Matrix on Burn Wounds
Acronym: Hyalomatrix
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision to not to proceed
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R14-090
Record Dates: First submitted 2015-01-28; First posted 2015-02-16 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyalomatrix (Active Comparator): Sterile, single use, flexible, and conformable wound dressing comprised of a derivative of hyaluronic acid which acts as a three dimensional regenerative matrix.
  Interventions: Device: Hyalomatrix
- Integra (Active Comparator): Sterile, single use, wound care dressing comprised of a porous matrix of cross-linked bovine tendon collagen and glycosaminoglycan
  Interventions: Device: Integra

INTERVENTIONS:
Device: Hyalomatrix
  Arms: Hyalomatrix
Device: Integra
  Arms: Integra

SUMMARY:
The purpose of this randomized, comparative study is to determine whether Hyalomatrix is as effective as IntegraTM Meshed Bilayer Wound Matrix when used in subjects who receive concurrent treatments with both products on their first and/or second degree burns located on both hands.

ELIGIBILITY:
Inclusion Criteria:

* Written consent must be obtained
* First and/or second degree burns on both hands
* Subject must be enrolled within 48 hours of the injury occurrence.

Exclusion Criteria:

* Subject is breastfeeding, pregnant, or has intentions of becoming pregnant during the course of their study participation.
* Subject has a prognosis that indicates unlikely survival past the study period.
* Subject's diagnosis indicates third degree burns.
* Subject suffers from burns sustained as a result of an electrical/chemical injury or by frostbite.
* Subject suffers from any inhalation-related burn trauma.
* Subject suffers from ongoing bone fractures.
* Subject has a known sensitivity to materials containing silicone, hyaluronan, bovine collagen, or chondroitin and/or derivatives of these products.
* Subject has received any treatment prior to study enrollment that may, in the opinion of the Investigator, affect the outcome of the study.
* Subject suffers from a medical condition that may impede wound healing, above any beyond that which would typically be expected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Wound Infection Rate | Up to 21 days
Number of days required for wound healing | Up to 21 days

SECONDARY OUTCOMES:
Range of Motion Scores | Up to 21 days
  Analysis of Range of Motion Scores
Physician Scores on Products Ease of Use | Up to 21 days
  Analysis of physician scores